CLINICAL TRIAL: NCT06416553
Title: Home-based Non-invasive Brain Stimulation in Combination With Lee Silverman Voice Treatment on Hypokinetic Dysarthria in Parkinson's Disease
Brief Title: Effect of Speech Therapy in Combination With Non-invasive Brain Stimulation on Speech of Patients With Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NU22J-04-00074
Record Dates: First submitted 2024-02-08; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A two parallel group, randomized, placebo controlled design will be used. Twenty PD patients will be stimulated for 4 weeks (20 sessions), stimulation will be combined with speech therapy . Other twenty PD patients will be stimulated with the same protocol using sham stimulation, sham stimulation will be combined with speech therapy.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD patients with real tDCS and speech therapy (Active Comparator): Patients will receive real tDCS during 4 weeks, 5 sessions per week. Altogether 20 sessions, each 20 minutes long. Stimulation is combined with Lee-Silverman voice treatment, 4 sessions per week. Altogether 16 sessions, each 1 hour long.
  Interventions: Device: Home-based transcranial direct current stimulation- real tDCS; Behavioral: Lee-Silverman voice treatment
- PD patients with sham tDCS and speech therapy (Sham Comparator): Patients will receive sham tDCS during 4 weeks, 5 sessions per week. Altogether 20 sessions, each 20 minutes long. Stimulation is combined with Lee-Silverman voice treatment, 4 sessions per week. Altogether 16 sessions, each 1 hour long.
  Interventions: Device: Home-based transcranial direct current stimulation- sham tDCS; Behavioral: Lee-Silverman voice treatment

INTERVENTIONS:
Device: Home-based transcranial direct current stimulation- real tDCS — Home-based transcranial direct current stimulation- anode over right STG, cathode over left STG, 2 mA stimulation with 1x1 tDCS mini-CT device by Soterix Medical
  Arms: PD patients with real tDCS and speech therapy
Device: Home-based transcranial direct current stimulation- sham tDCS — Home-based transcranial direct current stimulation- anode over right STG, cathode over left STG, sham stimulation with tDCS mini-CT device by Soterix Medical
  Arms: PD patients with sham tDCS and speech therapy
Behavioral: Lee-Silverman voice treatment — Remote Lee Silverman Voice Treatment (LSVT) delivered via telepractice by speech therapist. LSVT is a high-effort speech therapy that is primarily focused on improving speech loudness during 16 individual one-hour sessions in one month.

SUMMARY:
Up to 90% of patients with Parkinson's disease (PD) have hypokinetic dysarthria (HD) in the early phase of the illness. HD is characterized by a harsh breathy voice quality, reduced variability of pitch and loudness and imprecise articulation. This project investigates the novel combination of speech therapy and home-based non-invasive brain stimulation (tDCS) treatment in order to increase overall positive effects on HD in PD. Using a novel multimodal analysis approach based on functional magnetic resonance and acoustic signal processing, we will be able to monitor changes in different domains of speech, as well as associated changes in brain plasticity.

DETAILED DESCRIPTION:
Study will investigate the long-term effects of repeated (20) sessions of home-based tDCS as an add-on to well-established remote LSVT (i.e. the gold standard procedure for HD treatment) as compared to LSVT alone (coupled with sham stimulation) in patients with PD in their "on" dopaminergic condition without dyskinesias.

A two parallel-group, double-blinded, randomized, sham-stimulation-controlled design will be used. Forty PD patients will be randomized into two parallel groups by independent researcher by a computer-generated random number list, 20 subjects in each arm. Participants in the real tDCS group and the sham tDCS group will undergo a baseline assessment (V0), a follow-up assessment after four weeks of combined tDCS and LSVT treatments (V1) and another follow-up assessment 8 weeks after the baseline assessment (V2). Each visit will consist of EEG, speech tasks recording and speech evaluation by a speech therapist; MR scanning will be done at V0 and V1. Both groups will undergo the same speech therapy (LSVT) via telepractice as the gold standard treatment for HD, in combination with real or sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinically established PD (Postuma et al. 2016)

Exclusion Criteria:

* psychiatric disorders, including major depression, hallucinations
* any MRI-incompatible metal in the body
* epilepsy
* lack of cooperation
* presence of dementia

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in score of the 3F Test (the unabbreviated title- "the 3F Test Dysarthric Profile") | At baseline assessment (Visit- V0), after completion of 4 weeks of intervention (stimulation+ speech therapy) (Visit V1) and 4 weeks after completion of intervention (Visit V2)
  The 3F Test Dysarthric Profile enables clinicians to characterize a wide range of signs and symptoms of dysarthria. The minimum value of this scale is 0 (anarthria), the maximum value is 90 (no disorder). Higher scores of this scale mean better outcome. This test will be administrated by speech pathologist.

SECONDARY OUTCOMES:
Resting state fMRI | At baseline assessment (Visit- V0), after completion of 4 weeks of intervention (stimulation+ speech therapy) (V1) and 4 weeks after completion of intervention (V2)
  The effect of stimulation on the resting state networks will be studied using fMRI measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Central European Institute of Technology, Brno, Czechia